CLINICAL TRIAL: NCT03716297
Title: A Study of Some Aspects of Health in Special Youth Care: a Pilot Study
Brief Title: A Study of Some Aspects of Health in Special Youth Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Astrid Leenders, Principal Investigator, Vrije Universiteit Brussel
Other Study IDs: VrijeUB ALeenders
Record Dates: First submitted 2018-10-17; First posted 2018-10-23 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine some aspects of health in the special youth care. In this case it concerns the mental, social and physical and sporting health of the young people in the community institution De Kempen, Campus de Hutten. To examine these aspects of health, questionnaires will be used and participants will be asked to wear a SenseWear bracelet during their PE lessons. It is a pilot study that explores and tests the way in which certain things are best investigated in this setting. It examines how the practical side of such research should be carried out. It will also be investigated which obstacles, weaknesses and errors can be encountered when conducting such an investigation.

DETAILED DESCRIPTION:
This research is a quantitative cross-sectional study. Questionnaires will be taken from participants to measure mental, social and physical health. In addition, Sensewear bracelets will be used during the PE lessons of the participants to collect data (MET's and number of steps).

Three short questionnaires will be taken from the boys which measure the mental, social and physical health. Completing these questionnaires will take no longer than 10 minutes in total. The questionnaires will be filled in once by each participating individual at the start of the PE lesson.

During the PE class, the participants will receive a Sensewear bracelet in which the number of METs and the number of steps during the effort are measured. A distinction will also be made between the various sports during the PE lesson. Each participant will have to wear the Sensewear bracelet once during a single PE lesson.

It is an open research in which the participants are fully informed. The participants can voluntarily choose whether or not to participate in the study. The quantitative data collected from the questionnaires and Sensewear bracelets will then be used for de-finitive interpretation and decision making.

ELIGIBILITY:
Inclusion Criteria:

* For this research, data will only be collected from male participants with the age of 13 t.e.m. 18 years. These boys are in the (closed) Community institution De Kempen, Campus de Hutten.

Exclusion Criteria:

* For this research, no data will be collected from the young people on the other campus of the community institution. Campus de Markt is the open part of the community institution and the young people who live here are not the target group of the research.

Ages: 13 Years to 18 Years | Sex: Male
Age Groups: Child, Adult
Study Population: Male participants with the age of 13 t.e.m. 18 years who live in the (closed) Community institution De Kempen, Campus de Hutten.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The level of physical health in special youth care by using a questionnaire: The Physical Activity Questionnaire for Adolescents | 1 hour
  Use of a questionnaire (The Physical Activity Questionnaire for Adolescents) to assess physical health: there are 9 items in this questionnaire but only the first 8 items are used to calculate the total score. For the score of the first item you take the average of all the activities. On the other items the scores are between 1 and 5. To calculate the total score for this questionnaire, you have to calculate the average for all the 8 items. The final score is between 1 and 5 with 1 indicates low physical activity and 5 indicates high physical activity.
The level of mental health in special youth care by using a questionnaire: the Mental Health Inventory 5 | 1 hour
  Use of a questionnaire (Mental Health Inventory 5) to assess mental health: this questionnaire uses 5 questions to assess mental health. The score on each question is between 0 and 5. To calculate the total score of this questionnaire you have to add the scores of all the 5 questions and multiply by 4. The minimum sum score of a person is equal to 0 and the maximum score is equal to 100. The lower the score, the worse the psychological health of the person
The level of social health in special youth care by using a questionnaire: the Social Functioning Questionnaire | 1 hour
  Use of a questionnaire (the Social Functioning Questionnaire) to assess social health: The questionnaire consists of 8 items with 4 answer options each. The score of each item is between 0 and 3. The final score of the SFQ is calculated by adding the score of all items. The total score is then between 0 and 24, with a higher score indicating poorer social functioning.

SECONDARY OUTCOMES:
The level of physical activity during PE lessons in special youth care | 1 hour
  use of a sensewear bracelet

CONTACTS AND LOCATIONS:
Overall Officials: Evert Zinzen, Professor, Principal Investigator — Vrije Universiteit Brussel

IPD SHARING:
Plan to Share IPD: No